CLINICAL TRIAL: NCT06138834
Title: Effects of Y-6 Sublingual Tablets for Patients With Acute Ischemic Stroke: A Phase Ⅱ, Randomized, Double-blind, Double-dummy, Placebo-controlled Parallel Trial
Brief Title: EFfects of Y-6 SUblingual Tablets foR PaTients With AcUte Ischemic StRokE (FUTURE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YW2023-038-02
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Reperfusion
Keywords: Y-6; cilostazol; dexborneol; acute ischemic stroke; large vessel occlusion; reperfusion therapy; FUTURE
MeSH Terms: conditions — Ischemic Stroke | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dose Y-6 sublingual tablet group (Experimental): One Y-6 sublingual tablet (each tablet contains 25 mg Cilostazol and 6 mg Dexborneol), one placebo of Y-6 sublingual tablet (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol).
  Interventions: Drug: Low-dose Y-6 sublingual tablets
- High-dose Y-6 sublingual tablet group (Experimental): Two Y-6 sublingual tablets (each tablet contains 25 mg Cilostazol and 6 mg Dexborneol), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol).
  Interventions: Drug: High-dose Y-6 sublingual tablets
- Low-dose Cilostazol group (Experimental): Two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), one half Cilostazol tablet (each tablet contains 50 mg Cilostazol), and one half Cilostazol mimicry tablet(each tablet contains 0 mg Cilostazol).
  Interventions: Drug: Low-dose Cilostazol
- High-dose Cilostazol group (Experimental): Two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol tablet (each tablet contains 50 mg Cilostazol).
  Interventions: Drug: High-dose Cilostazol
- Placebo group (Placebo Comparator): Two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose Y-6 sublingual tablets — Take one Y-6 sublingual tablet (each tablet contains 25 mg Cilostazol and 6 mg Dexborneol), one placebo of Y-6 sublingual tablet (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol) for 28 days continuously.
  Arms: Low-dose Y-6 sublingual tablet group
Drug: High-dose Y-6 sublingual tablets — Take two Y-6 sublingual tablets (each tablet contains 25 mg Cilostazol and 6 mg Dexborneol), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol) for 28 days continuously.
  Arms: High-dose Y-6 sublingual tablet group
Drug: Low-dose Cilostazol — Take two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), one half Cilostazol tablet (each tablet contains 50 mg Cilostazol), and one half Cilostazol mimicry tablet(each tablet contains 0 mg Cilostazol) for 28 days continuously.
  Arms: Low-dose Cilostazol group
Drug: High-dose Cilostazol — Take two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol tablet (each tablet contains 50 mg Cilostazol) for 28 days continuously.
  Arms: High-dose Cilostazol group
Drug: Placebo — Take two tablets of placebo of Y-6 sublingual tablets (each tablet contains 0 mg Cilostazol and 0.06 mg Dexborneol to simulate the cool taste of Y-6 sublingual tablets when taken), and two halves Cilostazol mimicry tablets (each tablet contains 0 mg Cilostazol) for 28 days continuously.
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the efficacy of Y-6 sublingual tablets in improving microcirculation dysfunction and reducing thrombo-inflammation in patients who had AIS caused by LVO and received reperfusion therapy. Moreover, we expect to evaluate the safety of using Y-6 sublingual tablet in such study population.

DETAILED DESCRIPTION:
This study rationale is based on the following scheme: in patients with acute ischemic stroke caused by LVO, receiving reperfusion therapy may cause futile recanalization and thus lead to microcirculation dysfunction and thrombo-inflammation as consequences. Cilostazol has antiplatelet effects and BBB protection and Dexborneol has anti-inflammatory effects; therefore, the multi-component tablet may exert neuroprotective effects in terms of improving microcirculation dysfunction and reducing thrombo-inflammation in patients with AIS after reperfusion therapy.

The primary purpose of this study is to investigate the proportion of modified-Rankin scale (mRS) score recovered to 0~1 score at 90±7 days after randomization.

The follow-up duration is 3 months, and the visit schedule is as follows: Subjects enrolled based on randomization procedures will receive visits at screening/baseline period, 24 ± 2 hours, 7 ± 2 days, 28 + 3 days and 90 ± 7 days after randomization, and in case of any events.

ELIGIBILITY:
Inclusion Criteria:

* 35 years old ≤ Age ≤ 80 years old;
* Patients with acute ischemic stroke diagnosed within 24 hours of onset (time from onset to start of endovascular treatment);
* Patients with first stroke or mRS score 0-1 prior to this onset ;
* Patients with acute intracranial large vessel occlusion (LVO) confirmed by imaging examination, including occlusion of intracranial segments of internal carotid arteries, T-shaped bifurcation, MCA M1 and/or M2 segments and ACA A1 and/or A2 segments;
* ASPECTS score ≥ 6 when screening;
* 6<NIHSS score ≤ 25 after this onset;
* Patients who had the indications for mechanical thrombectomy and were scheduled for endovascular treatment;
* Patients or his/her legal representatives were able to understand and sign the informed consent.

Exclusion Criteria:

* Severe disorder of consciousness: NIHSS 1a consciousness level ≥2 points;
* Patients with definite history of intracranial hemorrhage, including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/external hematoma, etc. when screening;
* Patients with previously diagnosed intracranial tumor, arteriovenous malformation, or aneurysm when screening;
* Patients with bilateral LVO at anterior circulation or LVO at posterior circulation when screening;
* Patients with LVO of unknown or rare etiology, e.g., due to dissection, vasculitis, etc. when screening;
* Patients who have received treatment with tirofiban, warfarin, novel oral anticoagulants, argatroban, snake venom, defibrase, lumbrokinase or other defibrase therapy after onset, or platelet count <100×10^9/L;
* Patients with severe hepatic insufficiency or renal insufficiency and received dialysis for various reasons when screening (severe hepatic insufficiency was defined as ALT > 3 × ULN or AST >3 × ULN; severe renal insufficiency was defined as serum creatinine >3.0 mg/dl (265.2 μmol/L) or creatinine clearance < 30 ml/min);
* Patients with previously diagnosed hemorrhagic tendency (including but not limited to): with hereditary hemorrhagic disorders, such as hemophilia, when screening;
* Patients with refractory hypertension that is difficult to be controlled by medication (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg);
* Patients with history of major head trauma or stroke within 1 month prior to randomization;
* Patients who have received intracranial or spinal surgery within 3 months prior to randomization;
* Patients with history of major surgery or serious physical trauma within 1 month prior to randomization;
* Patients with previously diagnosed hemorrhagic retinopathy;
* Male subjects (or their mates) or female subjects who had planned to have a child during the whole study period and within 3 months after the end of the study period or were unwilling to use one or more non-drug contraceptive methods (e.g., complete abstinence, condoms, ligation, etc.) during the study period;
* Patients with contraindications to known contrast agents or other contrast agents; patients who are allergic to Cilostazol or Dexborneol;
* Patients who plan to receive other surgical or intervention therapy within 3 months, which might require discontinuation of the study drugs;
* Patients with life expectancy of less than 3 months due to advanced stage of comorbidity;
* Patients who have received treatment of investigational drugs or devices within previous 3 months;
* Other investigator-evaluated conditions which may influence the compliance of patients or where it is not suitable for patients to participate in this trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of mRS score recovered to 0~1 score | At 90±7 days after randomization
  The modified Rankin Scale (mRS) decreasing to 0~1 score. mRS Mainly measures patients' independent living ability, including physical function, activity ability and participation in daily life. A score of 0 on the mRS Scale indicates no symptoms and a score of 5 indicates severe disability.

SECONDARY OUTCOMES:
The mRS score at 90±7 days after randomization | At 90±7 days after randomization
  The modified Rankin Scale (mRS) decreasing to 0~1 score. mRS Mainly measures patients' independent living ability, including physical function, activity ability and participation in daily life. A score of 0 on the mRS Scale indicates no symptoms and a score of 5 indicates severe disability.
Changes of NIHSS score between baseline and at 24 ± 2 hours, 7 ± 2 days and 28 + 3 days after randomization | At 24 ± 2 hours, 7 ± 2 days and 28 + 3 days after randomization
  NIHSS score after reperfusion therapy within 2 hours changing compared with baseline NIHSS. The NIHSS score ranges from 0 to 42. The higher the score, the more severe the nerve damage.
Proportion of patients with early progression of stroke at 24 ± 2 hours after randomization | At 24 ± 2 hours after randomization
  Early progression of stroke was defined as: within 7 days after onset, compared to baseline, an increase of ≥ 2 points in NIHSS; or an increase of ≥ 1 point in limb hemiplegia; or an increase of ≥ 1 point in consciousness disorder, excluding those caused by intracranial hemorrhage and other non-stroke causes such as cardiac insufficiency, liver insufficiency, renal insufficiency, etc.
Proportion of patients with combined vascular events at 90 ± 7 days after randomization | At 90 ± 7 days after randomization
  Combined vascular events were defined as: symptomatic stroke, myocardial infarction and vascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD+MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Hussein HM, Georgiadis AL, Vazquez G, Miley JT, Memon MZ, Mohammad YM, Christoforidis GA, Tariq N, Qureshi AI. Occurrence and predictors of futile recanalization following endovascular treatment among patients with acute ischemic stroke: a multicenter study. AJNR Am J Neuroradiol. 2010 Mar;31(3):454-8. doi: 10.3174/ajnr.A2006. Epub 2010 Jan 14. PMID 20075087
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] van Horn N, Kniep H, Leischner H, McDonough R, Deb-Chatterji M, Broocks G, Thomalla G, Brekenfeld C, Fiehler J, Hanning U, Flottmann F. Predictors of poor clinical outcome despite complete reperfusion in acute ischemic stroke patients. J Neurointerv Surg. 2021 Jan;13(1):14-18. doi: 10.1136/neurintsurg-2020-015889. Epub 2020 May 15. PMID 32414889
- [Background] Casetta I, Fainardi E, Saia V, Pracucci G, Padroni M, Renieri L, Nencini P, Inzitari D, Morosetti D, Sallustio F, Vallone S, Bigliardi G, Zini A, Longo M, Francalanza I, Bracco S, Vallone IM, Tassi R, Bergui M, Naldi A, Saletti A, De Vito A, Gasparotti R, Magoni M, Castellan L, Serrati C, Menozzi R, Scoditti U, Causin F, Pieroni A, Puglielli E, Casalena A, Sanna A, Ruggiero M, Cordici F, Di Maggio L, Duc E, Cosottini M, Giannini N, Sanfilippo G, Zappoli F, Cavallini A, Cavasin N, Critelli A, Ciceri E, Plebani M, Cappellari M, Chiumarulo L, Petruzzellis M, Terrana A, Cariddi LP, Burdi N, Tinelli A, Auteri W, Silvagni U, Biraschi F, Nicolini E, Padolecchia R, Tassinari T, Filauri P, Sacco S, Pavia M, Invernizzi P, Nuzzi NP, Marcheselli S, Amista P, Russo M, Gallesio I, Craparo G, Mannino M, Mangiafico S, Toni D; Italian Registry of Endovascular Treatment in Acute Stroke. Endovascular Thrombectomy for Acute Ischemic Stroke Beyond 6 Hours From Onset: A Real-World Experience. Stroke. 2020 Jul;51(7):2051-2057. doi: 10.1161/STROKEAHA.119.027974. Epub 2020 Jun 17. PMID 32568647
- [Background] Berkhemer OA, Jansen IG, Beumer D, Fransen PS, van den Berg LA, Yoo AJ, Lingsma HF, Sprengers ME, Jenniskens SF, Lycklama A Nijeholt GJ, van Walderveen MA, van den Berg R, Bot JC, Beenen LF, Boers AM, Slump CH, Roos YB, van Oostenbrugge RJ, Dippel DW, van der Lugt A, van Zwam WH, Marquering HA, Majoie CB; MR CLEAN Investigators. Collateral Status on Baseline Computed Tomographic Angiography and Intra-Arterial Treatment Effect in Patients With Proximal Anterior Circulation Stroke. Stroke. 2016 Mar;47(3):768-76. doi: 10.1161/STROKEAHA.115.011788. Epub 2016 Jan 28. PMID 26903582
- [Background] Groot AE, Treurniet KM, Jansen IGH, Lingsma HF, Hinsenveld W, van de Graaf RA, Roozenbeek B, Willems HC, Schonewille WJ, Marquering HA, van den Berg R, Dippel DWJ, Majoie CBLM, Roos YBWEM, Coutinho JM; MR CLEAN Registry Investigators. Endovascular treatment in older adults with acute ischemic stroke in the MR CLEAN Registry. Neurology. 2020 Jul 14;95(2):e131-e139. doi: 10.1212/WNL.0000000000009764. Epub 2020 Jun 11. PMID 32527972
- [Background] Hussein HM, Saleem MA, Qureshi AI. Rates and predictors of futile recanalization in patients undergoing endovascular treatment in a multicenter clinical trial. Neuroradiology. 2018 May;60(5):557-563. doi: 10.1007/s00234-018-2016-2. Epub 2018 Mar 25. PMID 29574600
- [Background] Rubiera M, Garcia-Tornel A, Olive-Gadea M, Campos D, Requena M, Vert C, Pagola J, Rodriguez-Luna D, Muchada M, Boned S, Rodriguez-Villatoro N, Juega J, Deck M, Sanjuan E, Hernandez D, Pinana C, Tomasello A, Molina CA, Ribo M. Computed Tomography Perfusion After Thrombectomy: An Immediate Surrogate Marker of Outcome After Recanalization in Acute Stroke. Stroke. 2020 Jun;51(6):1736-1742. doi: 10.1161/STROKEAHA.120.029212. Epub 2020 May 14. PMID 32404034
- [Background] Ng FC, Coulton B, Chambers B, Thijs V. Persistently Elevated Microvascular Resistance Postrecanalization. Stroke. 2018 Oct;49(10):2512-2515. doi: 10.1161/STROKEAHA.118.021631. PMID 30355104
- [Background] Raja R, Rosenberg GA, Caprihan A. MRI measurements of Blood-Brain Barrier function in dementia: A review of recent studies. Neuropharmacology. 2018 May 15;134(Pt B):259-271. doi: 10.1016/j.neuropharm.2017.10.034. Epub 2017 Oct 28. PMID 29107626
- [Background] Bai R, Li Z, Sun C, Hsu YC, Liang H, Basser P. Feasibility of filter-exchange imaging (FEXI) in measuring different exchange processes in human brain. Neuroimage. 2020 Oct 1;219:117039. doi: 10.1016/j.neuroimage.2020.117039. Epub 2020 Jun 10. PMID 32534125
- [Derived] Wang Y, Qiu B, Guan L, Qu H, Pan Y, Huo X, Liu L, Miao Z, Li S, Li Z, Zhao X, Wang Y, Wang L, Liao X, Wang Y. EFfects of Y-6 SUblingual Tablets for PaTients with AcUte Ischemic StRokE (FUTURE): a phase II, randomised, double-blind, double-dummy, placebo-controlled, parallel trial. Stroke Vasc Neurol. 2025 Dec 23;10(6):793-799. doi: 10.1136/svn-2024-003666. PMID 40246318